CLINICAL TRIAL: NCT00002522
Title: HIGH-DOSE CYCLOPHOSPHAMIDE, ETOPOSIDE, AND CISPLATIN (CEP) WITH RESCUE BY AUTOLOGOUS BONE MARROW OR AUTOLOGOUS PERIPHERAL BLOOD STEM CELLS IN PATIENTS WITH RELAPSED OR REFRACTORY HODGKIN'S DISEASE
Brief Title: Combination Chemotherapy Followed by Bone Marrow or Peripheral Stem Cell Transplantation in Treating Patients With Relapsed or Refractory Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Temple University Bone Marrow Transplant Program, Temple University Health Systems
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000078283; TUHSC-2162; NCI-V93-0249
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Cisplatin; Cyclophosphamide; Etoposide; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: cyclophosphamide
Drug: etoposide
Procedure: autologous bone marrow transplantation
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation
Procedure: syngeneic bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with bone marrow or peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy followed by bone marrow or peripheral stem cell transplantation in treating patients with relapsed or refractory Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the curative potential of high-dose cyclophosphamide, etoposide, and cisplatin (CEP) followed by syngeneic or autologous bone marrow and/or autologous peripheral blood stem cell (PBSC) rescue in patients with relapsed or refractory stage I-IV Hodgkin's lymphoma.
* Determine the overall response rate and survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine the differences in the rate of engraftment, response, and survival of patients treated with bone marrow vs PBSC transplantation.
* Determine the response rate and survival of patients treated with late consolidative radiotherapy after recovery from transplantation.
* Determine the toxicity of late consolidative radiotherapy after recovery from transplantation in these patients.

OUTLINE: Syngeneic or autologous bone marrow and/or autologous peripheral blood stem cells (PBSC) are harvested. Syngeneic bone marrow transplantation is preferred for patients with a qualifying identical twin donor. Patients without a syngeneic donor who have a history of lymphomatous involvement of the bone marrow or are profoundly hypocellular undergo harvest of PBSC alone. Patients without a syngeneic donor who have no history of lymphomatous involvement of the bone marrow undergo harvest of autologous bone marrow or PBSC.

Patients receive conditioning comprising cyclophosphamide IV over 1 hour on days -6 to -3 and etoposide IV over 1 hour every 12 hours and cisplatin IV continuously on days -6 to -4. Bone marrow and/or PBSC are infused on day 0. (Patients requiring more than 25 bags of stem cells receive bone marrow transplantation on day 0 and PBSC transplantation on day 1.)

After recovery from transplantation, eligible patients receive consolidative radiotherapy to any site of prior bulk disease (greater than 5 cm) present at any time before transplantation and any site of disease present at the time of transplantation.

Patients are followed at 3, 6, and 12 months and then annually thereafter.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage I-IV Hodgkin's lymphoma
* Must have refractory or relapsed disease, defined by 1 of the following:

  * Failure to achieve a complete remission (CR) after 4 courses of conventional-dose front-line chemotherapy
  * Disease in second or greater remission

    * Patients should be encouraged to undergo transplantation prior to a third salvage regimen
    * Patients previously treated with multiple regimens considered on a case-by-case basis
* No chemoresistant disease, defined as active progression with tumor growth greater than 25% by volume during first-line chemotherapy

  * Patients who respond to second-line chemotherapy may be eligible
* Stable residual masses after conventional-dose chemotherapy not considered treatment failures

  * Active (refractory or relapsed) disease must be proven histologically or documented by gallium nitrate uptake
* Syngeneic marrow transplantation offered to patients with consenting identical twin donor
* No CNS involvement by lymphoma

PATIENT CHARACTERISTICS:

Age:

* 15 to 60 (selected patients up to age 70 may be eligible)

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 4,000/mm^3
* Absolute neutrophil count greater than 2,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL
* SGOT and SGPT less than 2 times upper limit of normal
* Albumin greater than 3.0 g/dL

Renal:

* Must meet 1 of the following criteria:

  * Creatinine less than 1.8 mg/dL
  * Creatinine clearance greater than 60 mL/min
  * BUN less than 20 mg/dL

Cardiovascular:

* Left ventricular ejection fraction at least 50%

Pulmonary:

* DLCO, FEV_1, and FVC greater than 50% of predicted OR
* Resting pO_2 greater than 70 mm Hg on room air

Other:

* HIV negative
* No severe neurologic or emotional disorders
* No active infection
* No other disease that would limit life expectancy
* Not pregnant
* Fertile patients must use effective contraception
* Adequate psychosocial support required

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-02; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth F. Mangan, MD, FACP, Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase - Temple Cancer Center, Philadelphia, Pennsylvania, United States